CLINICAL TRIAL: NCT02336204
Title: Effect of Alcohol Consumption and Nutritional Knowledge on Body Weight and Composition in a Group of Piacenza Students
Brief Title: Alcohol Consumption Relation With Nutritional Knowledge and Body Weight
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Filippo Rossi, researcher, Catholic University of the Sacred Heart
Other Study IDs: 24447/14
Record Dates: First submitted 2014-12-16; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The increase of overweight and obesity in young Italian people, nowadays showed by several epidemiological data, has been related to the misuse of alcohol and to a lack in nutritional knowledge.

Thus the aim of our study was to investigate if different nutritional knowledge from could affect body composition and drinking habits of a cohort of local young people.

104 healthy subjects (56 males and 54 females) were recruited using oral advertisements among the students of 18-19 years-old belonging to the Istituto Agrario and the Istituto alberghiero Raineri-Marcora of Piacenza. The subjects were asked to complete a questionnaire on alcohol consumption and another one related to nutritional knowledge. Then anthropometric data were measured: height, weight, waist and hips circumferences, waist-hips ratio and skinfolds were evaluated for each subject and body fat mass was calculated.

ELIGIBILITY:
Inclusion Criteria:

* students

Exclusion Criteria:

* pregnant or breast feeding
* vegan or vegetarian

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 104 healthy subjects (56 males and 54 females)
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
anthropometric measures | 1day
questionnaires on nutritional knowledge | 1 day